CLINICAL TRIAL: NCT01072448
Title: A 12-week Treatment, Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Assess the Efficacy and Safety of Once Daily Indacaterol in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: 12-week Efficacy of Indacaterol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2354
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Results first posted 2011-08-19 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; indacaterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Indacaterol 75 μg (Experimental): Patients inhaled indacaterol 75 μg once daily in the morning between 8:00 AM and 11:00 AM via a single-dose dry-powder inhaler (SDDPI) for 12 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 75 μg
- Placebo to indacaterol (Placebo Comparator): Patients inhaled placebo to indacaterol once daily in the morning between 8:00 AM and 11:00 AM via a single-dose dry-powder inhaler (SDDPI) for 12 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Placebo to indacaterol

INTERVENTIONS:
Drug: Indacaterol 75 μg — Indacaterol was supplied in powder filled capsules together with a single-dose dry-powder inhaler (SDDPI) device.
  Arms: Indacaterol 75 μg
Drug: Placebo to indacaterol — Placebo to indacaterol was supplied in powder filled capsules together with a single-dose dry-powder inhaler (SDDPI) device.
  Arms: Placebo to indacaterol

SUMMARY:
This 12-week study evaluated the efficacy and safety of indacaterol versus placebo.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of chronic obstructive pulmonary disease (COPD) (moderate-to-severe as classified by the Global Initiative for Chronic Obstructive Lung Disease [GOLD] Guidelines, 2008) and:

  * Smoking history of at least 10 pack-years
  * Post-bronchodilator forced expiratory volume in 1 second (FEV1) < 80% and ≥ 30% of the predicted normal value
  * Post-bronchodilator FEV1/FVC (forced vital capacity) < 70%

Exclusion criteria:

* Patients who have had a COPD exacerbation requiring systemic corticosteroids and/or antibiotics and/or hospitalization in the 6 weeks prior to screening
* Patients who have had a respiratory tract infection within 6 weeks prior to screening
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Any patient with lung cancer or a history of lung cancer
* Patients with a history of certain cardiovascular co-morbid conditions Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (60):
- United States (60):
  - Novartis Investigator Site, Peoria, Arizona
  - Novartis Investigator Site, Pine Bluff, Arkansas
  - Novartis Investigator Site, Buena Park, California
  - Novartis Investigator Site, Encinitas, California
  - Novartis Investigator Site, Fountain Valley, California
  - Novartis Investigator Site, Los Angeles, California
  - Novartis Investigator Site, San Diego, California
  - Novartis Investigator Site, Temecula, California
  - Novartis Investigator Site, Torrance, California
  - Novartis Investigator Site, Walnut Creek, California
  - Novartis Investigator Site, Wheat Ridge, Colorado
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigator Site, Couer D'Alene, Idaho
  - Novartis Investigator Site, Champaign, Illinois
  - Novartis Investigator Site, Downers Grove, Illinois
  - Novartis Investigative Site, River Forest, Illinois
  - Novartis Investigator Site, Skokie, Illinois
  - Novartis Investigator Site, Springfield, Illinois
  - Novartis Investigative site, Lexington, Kentucky
  - Novartis Investigator Site, Covington, Louisiana
  - Novartis Investigator Site, Metaire, Louisiana
  - Novartis Investigative Site, Bangor, Maine
  - Novartis Investigative Site, Columbia, Maryland
  - Novartis Investigative Site, Clarkston, Michigan
  - Novartis Investigative Site, Flint, Michigan
  - Novartis Investigative Site, Livonia, Michigan
  - Novartis Investigative Site, Edina, Minnesota
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Plymouth, Minnesota
  - Novartis Investigator Site, Florissant, Missouri
  - Novartis Investigator Site, Ozark, Missouri
  - Novartis Investigator Site, St Louis, Missouri
  - Novartis Investigative Site, Missoula, Montana
  - Novartis Investigator Site, Bellevue, Nebraska
  - Novartis Investigator Site, Lincoln, Nebraska
  - Novartis Investigator Site, Omaha, Nebraska
  - Novartis Investigator Site, Henderson, Nevada
  - Novartis Investigator Site, Pahrump, Nevada
  - Novartis Investigative Site, New Brunswick, New Jersey
  - Novartis Investigative Site, Ocean City, New Jersey
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Salisbury, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigator Site, Medford, Oregon
  - Novartis Investigative Site, Beaver, Pennsylvania
  - Novartis Investigative Site, Erie, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Gaffney, South Carolina
  - Novartis Investigative site, Greer, South Carolina
  - Novartis Investigative Site, Seneca, South Carolina
  - Novartis Investigative Site, Johnson City, Tennessee
  - Novartis Investigator Site, Corsicana, Texas
  - Novartis Investigator Site, Fort Worth, Texas
  - Novartis Investigator Site, Salt Lake City, Utah
  - Novartis Investigator Site, Abingdon, Virginia
  - Novartis Investigative Site, Newport News, Virginia
  - Novartis Investigator Site, Tacoma, Washington

REFERENCES:
- [Derived] Gotfried MH, Kerwin EM, Lawrence D, Lassen C, Kramer B. Efficacy of indacaterol 75 mug once-daily on dyspnea and health status: results of two double-blind, placebo-controlled 12-week studies. COPD. 2012 Dec;9(6):629-36. doi: 10.3109/15412555.2012.729623. Epub 2012 Sep 28. PMID 23020650
- [Derived] Kerwin EM, Gotfried MH, Lawrence D, Lassen C, Kramer B. Efficacy and tolerability of indacaterol 75 mug once daily in patients aged >/=40 years with chronic obstructive pulmonary disease: results from 2 double-blind, placebo-controlled 12-week studies. Clin Ther. 2011 Dec;33(12):1974-84. doi: 10.1016/j.clinthera.2011.11.009. PMID 22177371

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indacaterol 75 μg | Placebo to Indacaterol
Started | 163 | 160
Completed | 144 | 130
Not Completed | 19 | 30
Not completed — Adverse Event | 9 | 10
Not completed — Subject withdrew consent | 4 | 9
Not completed — Protocol deviation | 3 | 4
Not completed — Abnormal test procedure result(s) | 1 | 0
Not completed — Unsatisfactory therapeutic effect | 1 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Abnormal laboratory value(s) | 0 | 1
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 75 μg | Placebo to Indacaterol | Total
Number analyzed (Participants) | 163 | 160 | 323
Age Continuous [Mean (Standard Deviation); unit: years] | 64.0 (8.29) | 64.1 (9.43) | 64.0 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 73 | 147
  Male | 89 | 87 | 176

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) 24 Hours Post-dose at the End of the Study (Week 12 + 1 Day, Day 85)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose at the end of treatment. The analysis included baseline FEV1, FEV1 pre-dose and 10-15 minutes post-dose of albuterol during screening, and FEV1 pre-dose and 50-70 minutes post-dose of ipratropium during screening as covariates.
Time Frame: 24 hours post-dose at the end of the study (Week 12 + 1 day, Day 85)
Population: Full analysis set: All randomized patients who received at least 1 dose of study drug, last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 75 μg | Placebo to Indacaterol
Number analyzed (Participants) | 149 | 148
Liters | 1.38 (0.013) | 1.26 (0.013)

2. Secondary Outcome: Transition Dyspnea Index (TDI) Total Score at the End of the Study (Week 12, Day 84)
Description: An independent (where feasible), trained assessor interviewed the patient and rated the degree of impairment due to dyspnea on a scale from -3 (major deterioration) to 3 (major improvement) on 3 domains (functional impairment, magnitude of task, and magnitude of effort) in comparison with baseline. A total score of the 3 domains ranged from -9 to 9; minus scores indicate deterioration. The analysis included baseline dyspnea index, FEV1 pre-dose and 10-15 minutes post-dose of albuterol during screening, and FEV1 pre-dose and 50-70 minutes post-dose of ipratropium during screening as covariates.
Time Frame: End of the study (Week 12, Day 84)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Indacaterol 75 μg | Placebo to Indacaterol
Number analyzed (Participants) | 150 | 150
Units on a scale | 1.34 (0.284) | 0.11 (0.287)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The safety set, included all patients who received at least one dose of study drug.
Arm/Group | Indacaterol 75 μg | Placebo to Indacaterol
Serious Adverse Events (participants affected / at risk) | 4/163 | 9/160
Other Adverse Events (participants affected / at risk) | 29/163 | 23/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 75 μg (N=163) | Placebo to Indacaterol (N=160)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 75 μg (N=163) | Placebo to Indacaterol (N=160)
Urinary tract infection (Infections and infestations) | 9 | 2
Headache (Nervous system disorders) | 9 | 6
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 14 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.